CLINICAL TRIAL: NCT04402632
Title: A Study of the Embolization of the Middle Meningeal Artery With ONYX™ Liquid Embolic System In the Treatment of Subacute and Chronic Subdural HEmatoma (EMBOLISE)
Brief Title: Embolization of the Middle Meningeal Artery With ONYX™ Liquid Embolic System for Subacute and Chronic Subdural Hematoma
Acronym: EMBOLISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Neurovascular Clinical Affairs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: MDT19027ONYX
Record Dates: First submitted 2020-05-18; First posted 2020-05-27 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Subdural Hematoma
MeSH Terms: conditions — Hematoma, Subdural | interventions — Embolization, Therapeutic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Surgery Cohort: Control Arm (Active Comparator)
  Interventions: Procedure: Surgical Management
- Surgery Cohort: Treatment Arm (Experimental)
  Interventions: Device: Onyx™ Liquid Embolic System (LES) Embolization; Procedure: Surgical Management
- Observational Cohort: Control Arm (Active Comparator)
  Interventions: Other: Observation Only
- Observational Cohort: Treatment Arm (Experimental)
  Interventions: Device: Onyx™ Liquid Embolic System (LES) Embolization

INTERVENTIONS:
Procedure: Surgical Management — Surgical Evacuation of the Subdural Hematoma (SDH) (Control)
  Arms: Surgery Cohort: Control Arm
Device: Onyx™ Liquid Embolic System (LES) Embolization — Onyx™ LES Embolization of the Subdural Hematoma (SDH)
  Arms: Surgery Cohort: Treatment Arm
Other: Observation Only — Medical Management (Control)
  Arms: Observational Cohort: Control Arm
Device: Onyx™ Liquid Embolic System (LES) Embolization — Onyx™ LES Embolization of the Subdural Hematoma (SDH)
  Arms: Observational Cohort: Treatment Arm
Procedure: Surgical Management — Surgical Evacuation of the Subdural Hematoma (SDH)
  Arms: Surgery Cohort: Treatment Arm

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of embolization of the middle meningeal artery (MMA) using the Onyx™ Liquid Embolic System (LES) for treatment of symptomatic subacute or chronic subdural hematoma (SDH)

ELIGIBILITY:
Inclusion Criteria:

* Pre-morbid Modified Rankin Score ≤3
* Confirmed diagnosis of subacute or chronic subdural hematoma
* Completed informed consent
* Meets criteria for Surgery or Observation Cohort

Exclusion Criteria:

* Life expectancy <1 year
* Unable to complete follow-up
* Pregnant, lactating, or has a positive pregnancy test at time of admission
* Diagnosed with acute SDH
* Potentially dangerous anatomic variations leading to increased procedural risk or unsafe access for MMA embolization
* Pre-randomized Markwalder Grading Scale score ≥ 3
* Unmanaged, uncontrolled bleeding disorders/blood diathesis
* Presumed septic embolus, or suspicion of microbial superinfection
* Known active COVID-19 infection
* CT or MRI evidence of intra-cranial tumor or mass lesion Contraindication to angiography
* Participation in another clinical trial
* Contraindicated for the use of Onyx™ LES
* Cannot be taken off corticosteroids (intended to treat subacute or chronic SDH) for at least 90 days post-randomization

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2025-04-03 (Actual)

PRIMARY OUTCOMES:
Rate of hematoma recurrence/progression requiring surgical drainage OR poor clinical outcome at 90 days, OR clinical deterioration at 90 days compared to baseline | 90 days post-procedure

SECONDARY OUTCOMES:
Non-inferiority assessment of Onyx™ LES embolization treatment compared to standard of care based on change in Modified Rankin Scale Score | 90 days post-procedure
Effectiveness: Incidence of hospital readmissions | 90 days post-procedure
Effectiveness: Change in hematoma volume based on CT/MRI imaging | 90 days post-procedure
Effectiveness: Change in hematoma thickness per CT/MRI imaging | 90 days post-procedure
Effectiveness: Change in midline shift based on CT/MRI imaging | 90 days post-procedure
Safety: Incidence of device-related serious adverse events | 30 days post-procedure
Safety: Incidence of procedure-related serious adverse events | 30 days post-procedure
Safety: Incidence of neurological death | 90 days and 180 days post-procedure
Safety: Incidence of device-related adverse events | 90 days and 180 days post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jared Knopman, MD, Principal Investigator — New York-Presbyterian Hospital/Weill Cornell Medical Center; Jason Davies, MD, Principal Investigator — Buffalo General Medical Center
Locations (49):
- United States (49):
  - University of Alabama at Birmingham (UAB) Hospital, Birmingham, Alabama
  - Carondelet St. Joseph's Hospital, Tucson, Arizona
  - University of California Irvine Medical Center, Irvine, California
  - USC - Keck School of Medicine, Los Angeles, California
  - Huntington Memorial Hospital, Pasadena, California
  - UCSD Medical Center, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - University of California San Francisco Medical Center, San Francisco, California
  - Providence Little Company of Mary Medical Center, Torrance, California
  - University of Colorado Denver School of Medicine, Aurora, Colorado
  - UF Health Heart and Vascular Hospital, Gainesville, Florida
  - Memorial Regional Hospital, Hollywood, Florida
  - Baptist Medical Center Jacksonville, Jacksonville, Florida
  - Jackson Memorial Hospital, Miami, Florida
  - Orlando Regional Medical Center Orlando Health, Orlando, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Ascension Saint Vincent Hospital, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kentucky Albert B Chandler Hospital, Lexington, Kentucky
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - McLaren Flint Hospital, Flint, Michigan
  - Corewell Health, Grand Rapids, Michigan
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Albany Medical Center, Albany, New York
  - Buffalo General Medical Center, Buffalo, New York
  - North Shore University Hospital, Manhasset, New York
  - The Mount Sinai Hospital, New York, New York
  - New York-Presbyterian Hospital/Weill Cornell Medical Center, New York, New York
  - Westchester Medical Center, Valhalla, New York
  - Atrium Health's Carolinas Medical Center, Charlotte, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University/Wexner Medical Center, Columbus, Ohio
  - ProMedica Toledo Hospital, Toledo, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Oregon Health & Science University Hospital, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - University of Pittsburgh Medical Center UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Prisma Health, Greenville, South Carolina
  - Valley Baptist Medical Center, Harlingen, Texas
  - Memorial Hermann-Texas Medical Center, Houston, Texas
  - Baylor Scott & White Medical Center - Temple, Temple, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - Harborview Medical Center, Seattle, Washington
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be available

REFERENCES:
- [Derived] Kniep H, Gellissen S, Bechstein M, Meyer L, Broocks G, Heitkamp C, Winkelmeier L, Flottmann F, Geest V, Hanning U, Thaler C, Bester M, Davies JM, Knopman J, Mokin M, Hassan AE, Harbaugh RE, Khalessi A, Siddiqui AH, Gross BA, Grandhi R, Tarpley J, Sivakumar W, Bain M, Crowley RW, Link TW, Fraser JF, Levitt MR, Chen PR, Hanel RA, Bernard JD, Jumaa M, Youssef P, Cress MC, Chaudry MI, Shakir HJ, Lesley WS, Billingsley J, Jones J, Koch MJ, Paul AR, Mack WJ, Osbun JW, Dlouhy K, Grossberg JA, Kellner CP, Sahlein DH, Santarelli J, Schirmer CM, Singer J, Liu JJ, Majjhoo AQ, Wolfe T, Patel NV, Roark C, Fiehler J; EMBOLISE Investigators. Middle Meningeal Artery Embolization for Subdural Hematoma: CT/MRI End Points of the EMBOLISE Trial. Radiology. 2026 Jan;318(1):e251746. doi: 10.1148/radiol.251746. PMID 41591252
- [Derived] Davies JM, Knopman J, Mokin M, Hassan AE, Harbaugh RE, Khalessi A, Fiehler J, Gross BA, Grandhi R, Tarpley J, Sivakumar W, Bain M, Crowley RW, Link TW, Fraser JF, Levitt MR, Chen PR, Hanel RA, Bernard JD, Jumaa M, Youssef P, Cress MC, Chaudry MI, Shakir HJ, Lesley WS, Billingsley J, Jones J, Koch MJ, Paul AR, Mack WJ, Osbun JW, Dlouhy K, Grossberg JA, Kellner CP, Sahlein DH, Santarelli J, Schirmer CM, Singer J, Liu JJ, Majjhoo AQ, Wolfe T, Patel NV, Roark C, Siddiqui AH; EMBOLISE Investigators. Adjunctive Middle Meningeal Artery Embolization for Subdural Hematoma. N Engl J Med. 2024 Nov 21;391(20):1890-1900. doi: 10.1056/NEJMoa2313472. PMID 39565988